CLINICAL TRIAL: NCT06273527
Title: Enhancing Transdiagnostic Mechanisms of Cognitive Dyscontrol
Brief Title: Enhancing Transdiagnostic Mechanisms of Cognitive Dyscontrol (R33)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jessica Bomyea, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 808681
Record Dates: First submitted 2024-01-31; First posted 2024-02-22 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Anxiety Disorders; Depression; Post Traumatic Stress Disorder
MeSH Terms: conditions — Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic | interventions — cogent db

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COGENT - Cognitive Training Intervention Program (Experimental): Computer-administered cognitive training program. COGENT is a modified working memory capacity task designed to train cognitive functioning. COGENT was designed to contain high interference across trials. By requiring repeated practice with utilization of interference control across trials, COGENT is thought to enhance plasticity of cognitive systems and improve performance. That is, training is based on the premise that learning-based neural changes will occur via repeated exposure to a task demanding cognitive control resources
  Interventions: Behavioral: COGENT
- Non-Training Program (Sham Comparator): The non-training condition requires participants to complete a similar computer task for the same length of time. The non-training is a modified working memory capacity task designed to be inert. The non-training condition was designed to contain relatively less interference demands across trials.
  Interventions: Other: Sham Program

INTERVENTIONS:
Behavioral: COGENT — COGENT is based on a working memory capacity task, which requires individuals to memorize stimuli while simultaneously completing a secondary puzzle task.
  Arms: COGENT - Cognitive Training Intervention Program
Other: Sham Program — The Sham Program will be a similar task which researchers think will be less effective in training thinking skills.
  Arms: Non-Training Program

SUMMARY:
The proposed project aims to test the cognitive and neural effects of a cognitive training in a sample of individuals seeking treatment for anxiety, depression, or traumatic stress symptoms. Participants will be randomly assigned to one of two groups. Group 1 will receive a computer-based program that is designed as a cognitive training intervention and Group 2 will receive a similar computer-based exercise that researchers think will be less effective in training thinking skills (also known as a control or sham condition). Participants will be compared on cognitive performance and brain response during cognitive tasks from baseline to post-treatment.

DETAILED DESCRIPTION:
Mood, anxiety, and traumatic stress disorders are common psychiatric conditions - affecting over 40 million U.S. adults - and are leading causes of disability worldwide. People with these conditions are commonly plagued by difficulty controlling distressing personal thoughts and memories, collectively referred to as repetitive negative thinking symptoms. Models suggest that repetitive negative thinking is driven by executive functioning deficits, such that cognitive resources are insufficient to downregulate unwanted thoughts. Executive functioning deficits could be a promising treatment target but are not typically addressed with existing interventions. The long-term goal advanced by this project is to develop effective, mechanistic cognitive training programs that can improve cognition and reduce symptoms associated with mood, anxiety, and traumatic stress disorders. The objectives of this proposal is to evaluate the cognitive effects of the optimized computer-based cognitive training intervention relative to a sham training program (ST). The central hypothesis is that the cognitive training intervention will enhance executive functioning and will lead to a reduction of repetitive negative thinking in mood, anxiety, and traumatic stress disorders. The project will randomize participants with depression, anxiety, and/or traumatic stress disorders to a cognitive training intervention program or a sham training program. The investigators will examine executive functioning change with cognitive task performance and functional neuroimaging assessments.

ELIGIBILITY:
Inclusion Criteria:

* age 21-55
* fluent in English
* diagnosis of mood, anxiety, or traumatic stress disorder
* clinically elevated repetitive negative thinking
* outpatient status
* 6-week stability if taking selective serotonin reuptake inhibitor (SSRI) medications

Exclusion Criteria:

* past year diagnosis of severe alcohol or moderate or greater substance use disorder
* lifetime history of psychotic or bipolar I disorder
* acute suicidality necessitating immediate clinical intervention
* neurodegenerative or neurodevelopmental disorders
* history of moderate or severe traumatic brain injury or other known neurological condition
* sensory deficits that would preclude completing tasks
* conditions unsafe for completing MRI scanning (e.g., metal in body)
* current pregnancy
* currently receiving psychosocial treatment
* currently receiving psychiatric pharmacotherapy, except SSRIs

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive performance | Baseline, Week 4, Week 8, Week 16
  Span Working Memory Score. Scores are calculated based on memory accuracy total points across all trials, with higher scores indicating better performance. This change is expected to be significantly higher for the COGENT group than the Sham group.

SECONDARY OUTCOMES:
Reading Span Blood Oxygen Level Dependent (BOLD) Response | Baseline, Week 4
  Functional Magnetic Resonance Imaging (fMRI) Reading span working memory capacity task while undergoing functional MRI. Neural activation to task condition is measured using % signal change (0-100) with higher scores indicating greater activation.
Neuropsychological Performance | Baseline, Week 4, Week 8, Week 16
  Change from baseline in neuropsychological performance as measured by a composite of the following tests Flanker Inhibitory Control and Attention Test, Picture Sequence Memory Test, List Sorting Working Memory Test, Oral Reading Recognition Test, Dimensional Change Card Sort Test, Pattern Comparison Processing Speed Test, Picture Vocabulary Test (measured at baseline and week 4) and Matrix Reasoning, Digit Span, Trail Making Test, Digit Symbol Matching.
Repetitive Negative Thinking (RNT) | Baseline, Week 4,Week 8, Week 16
  Change from baseline in RNT as measured by a composite of the Ruminative Response Scale (RRS), Penn State Worry Questionnaire (PSWQ), the Repetitive Negative Thinking Questionnaire-10 (RTQ-10) and the Perseverative Thinking Questionnaire (PTQ).
  The total score for the RRS ranges from 22 to 88, with higher scores indicating higher degrees of ruminative symptoms.
  The total score for the PSWQ ranges from 16 to 80, with higher scores indicating higher worry.
  The total score for the RTQ-10 ranges from 10 to 50, with higher scores indicating higher repetitive thinking.
  The total score for the PTQ ranges from 0 to 60, with higher scores indicating higher repetitive negative thinking. Scores of each characteristic of RNT can also be obtained.

OTHER OUTCOMES:
Disability | Baseline, Week 4,Week 8, Week 16
  Change from baseline in disability across six domains, understanding and communicating, getting around, self-care, getting along with people, life activities, and participation in society as measured by the World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0).
  A simple score for the WHODAS 2.0 ranges from 36-180 with higher scores indicating the degree of functional limitations. An item-response-theory based score can also be obtained by summing the recoded item scores within each of the six domains, summing the domains, and converting the summary score into a metric ranging from 0 to 100, with higher scores indicating higher disability.
Suicide Cognitions | Baseline, Week 4,Week 8, Week 16
  Change from baseline in suicide-related beliefs as measures by the Suicide Cognitions Scale-Revised (SCS-R). The total score ranges from 0 to 64, with higher scores indicating higher severity of suicidal cognitions.
Mood and Emotions | Baseline, Week 4,Week 8, Week 16
  Changes from baseline in mood and emotions as measured by the Positive and Negative Affect Schedule (PANAS).There are two scores calculated, one for positive affect and one for negative affect. The total score for positive affect ranges from 10 to 50. The total score for negative affect ranges from 11 to 55.
Self-reported attention | Baseline, Week 4,Week 8, Week 16
  Change from baseline in attention focusing and attention shifting as measured by the Attention Control Questionnaire. The total score ranges from 20 to 80, with higher scores indicating higher levels of attention control.
Anxiety Symptoms | Baseline, Week 4, Week 8, Week 16
  Change from baseline in anxiety symptoms as measured by General Anxiety Disorder 7 (GAD-7). The total score ranges from 0-21. With higher scores indicating higher levels of anxiety symptoms.
Symptoms of Depression | Baseline, Week 4, Week 8, Week 16
  Change from baseline in symptoms of depression as measured by the PhenX Depression-Quick Inventory of Depressive Symptoms (QUIDS). The total score ranges from 0-27, with higher scores indicating higher depressive symptoms.
PTSD Symptoms | Baseline, Week 4, Week 8, Week 16
  Change from baseline in PTSD symptoms as measured by PTSD Checklist for DSM-5 (PCL-5).The total score ranges from 0-80, with higher scores indicating higher severity.

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No